CLINICAL TRIAL: NCT02068820
Title: Detection of Sentinel Lymph Nodes in Patients With Endometrial Cancer Undergoing Robotic-Assisted Staging: Comparison of Isosulfan Blue (ISB) and Indocyanine Green Dyes (ICG) With Fluorescence Imaging
Brief Title: Detection of SLN in Patients With Endometrial Cancer Undergoing Robotic Assisted Staging: Comparison of ISB and ICG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AdventHealth (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SLN Mapping
Record Dates: First submitted 2014-02-14; First posted 2014-02-21 (Estimated); Results first posted 2019-09-10 (Actual); Last update posted 2019-09-10 (Actual); Status verified 2019-08

CONDITIONS: Endometrial Cancer
Keywords: Sentinel lymph nodes; da Vinci; Firefly; Sentinel lymph node mapping; Fluorescence Imaging; SLN; SLN mapping
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ISB dye, standard white light (Active Comparator): SLN mapping utilizing da Vinci surgical system with Isosulfan Blue (ISB) dye and standard white light imaging.
  Interventions: Device: ISB dye and standard white light imaging
- ICG dye, FireFly fluorescence imaging (Experimental): SLN mapping utilizing da Vinci surgical system with ISB dye and standard white light first, and then additionally, Indocyanine Green (ICG) dye and FireFly fluorescence imaging.
  Interventions: Device: ISB dye and standard white light imaging; Device: ICG dye and FireFly fluorescence imaging

INTERVENTIONS:
Device: ISB dye and standard white light imaging — Sentinel lymph node mapping utilizing the da Vinci surgical system and ISB dye with standard white light imaging.
  Other Names: Isosulfan Blue dye
Device: ICG dye and FireFly fluorescence imaging — Sentinel lymph node mapping utilizing the da Vinci surgical system with ICG dye and FireFly fluorescence imaging.
  Other Names: Indocyanine green dye
  Arms: ICG dye, FireFly fluorescence imaging

SUMMARY:
The investigators hypothesis is that if sensitivity and specificity are found to be significantly higher than the current reports with Technesium-99 and ISB colorimetric dye, SLN biopsies might allow omission of full lymphadenectomy in lower-risk cases, thereby limiting peri-operative morbidity. SLN biopsies might also improve the detection of metastatic disease, essentially lowering the recognized false-negative rate of standard lymphadenectomy analyzed by routine H&E pathologic analysis.

DETAILED DESCRIPTION:
The study objective is to compare two sentinel lymph node detection technologies [fluorescence imaging and Indocyanine Green (ICG) dye verses standard laparoscopic colorimetric analysis using Isosulfan Blue (ISB) dye] for sensitivity and specificity of detecting metastatic disease in pelvic lymph nodes of women with endometrial cancer undergoing robotic-assisted laparoscopic hysterectomy and lymphadenectomy. The following three specific aims would be addressed in this research proposal:

Specific Aim 1: To determine the ability of mapping bilaterally pelvic SLN in women with endometrial cancer undergoing robotic-assisted laparoscopic staging comparing two different methods (i.e., comparing the combination of colorimetric analysis-ISB dye + fluorescence imaging-ICG dye vs. colorimetric analysis-ISB dye alone).

Specific Aim 2: To estimate the negative predictive value (NPV) of pelvic SLN in endometrial cancer with respect to predicting nodal metastasis.

Specific Aim 3: To evaluate the ability of sentinel lymph nodes to increase the detection of metastatic disease through ultra-sectioning and immuno-histochemical (IHC) staining by comparing IHC results and standard hematoxylin and eosin (H&E) results.

ELIGIBILITY:
Inclusion Criteria:

1. The patient must be ≥18 and ≤85 years of age.
2. The patient must be female.
3. The patient must be willing and able to provide informed consent.
4. The patient is willing and able to comply with the study protocol.
5. The patient has endometrial cancer and is scheduled for robotic hysterectomy and lymphadenectomy.
6. The patient agrees to follow-up examinations out to 6-weeks post-treatment

Exclusion Criteria:

1. The patient is not a candidate for robotic assisted hysterectomy and lymphadenectomy.
2. The patient has known or suspected allergies to iodine, ICG or ISB.
3. The patient has hepatic dysfunction confirmed by elevated liver function studies (i.e., hepatic enzyme SGOT, SGPT or Bilirubin > 2 x normal (based on reference values from the laboratory used by the patient)

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2012-09; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Holloway, MD, Principal Investigator — Florida Hospital Gynecologic Oncology
Locations (1):
- Florida Hospital Gynecologic Oncology, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ISB Dye, Standard White Light | ICG Dye, FireFly Fluorescence Imaging
Started | 20 | 180
Completed | 20 | 180
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ISB Dye, Standard White Light | ICG Dye, FireFly Fluorescence Imaging | Total
Number analyzed (Participants) | 20 | 180 | 200
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 79 | 86
  >=65 years | 13 | 101 | 114
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 180 | 200
  Male | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20 | 180 | 200
Age [Median (Standard Deviation); unit: years] | 66.0 (6.7) | 64.4 (8.6) | 64.5 (8.4)

OUTCOME MEASURES:

1. Primary Outcome: Number of Pelvic Sentinel Lymph Nodes (SLN) in Endometrial Cancer Patients Detected by Either ICG and/or ISB Dyes.
Time Frame: through 6 weeks post-operative
Population: The ISB dye alone group (n=20) and the ICG group (n=180) are combined, because both groups received the ISB dye.
Measure: Mean (Standard Deviation); unit: nodes
Arm/Group | ISB Dye, Standard White Light | ICG Dye, FireFly Fluorescence Imaging
Number analyzed (Participants) | 200 | 180
nodes | 1.25 (.901) | 2.03 (.720)

2. Secondary Outcome: Negative Predictive Value (NPV) of Pelvic SLN in Endometrial Cancer in Relation to the Number of Nodes With Metastasis.
Description: The standard definition for negative predictive value was used to calculate NPV. There was one false negative SLN in this study, 39 true positive sentinel lymph nodes, and 140 negative pelvic metastatic patients.
  NPV = 140/141=99.3%
Time Frame: through 6 weeks post-operative
Population: Comparison of metastatic disease (yes or no) with ICG dye node detection (yes or no)
Measure: Count of Participants; unit: Participants
Groups:
- ICG Negative: Experimental subjects with Indocyanine Green (ICG) negative test results
- ICG Positive: Experimental subjects with Indocyanine Green (ICG) positive test results
Arm/Group | ICG Negative | ICG Positive
Number analyzed (Participants) | 141 | 39
Participants
  Metastatic Disease | 1 | 39
  Non Metastatic Disease | 140 | 0

3. Other Pre Specified Outcome: Number of Pelvic Sentinal Lymph Nodal Metastasis in Regard to Staining by Immunohistochemical (IHC) Staining in Comparison to Standard Hematoxylin and Eosin (H&E).
Description: Of the 127 positive nodes with pathology information, the percentage of each type of node will be summarized by the staining method. Statistical testing of the individual staining methods compared to both will be computed using Chi-square test of independence.
Time Frame: through 6 weeks post-operative
Population: These are positive sentinel lymph nodes
Measure: Number; unit: nodes
Units Other Than Participants: Nodes
Groups:
- IHC Only: Positive node identified with IHC dye only
- H&E Only: Positive node identified with H&E only
- Both IHC and H&E: Positive node identified with both IHC and H&E dye
Arm/Group | IHC Only | H&E Only | Both IHC and H&E
Number analyzed (Participants) | NA | NA | NA
Number analyzed (Nodes) | 18 | 91 | 18
nodes
  Sentinel Nodes | 16 | 31 | 16
  Pelvic Nodes Only | 1 | 36 | 2
  Aortic | 1 | 14 | 0
  Infrarenal | 0 | 10 | 0

ADVERSE EVENTS:
Time Frame: Post-op follow up 6 weeks
Groups:
- ISB Only Adverse Events: ISB only Adverse Events categories reported during post-op follow up 6 weeks
- ICG Adverse Events: ICG Adverse Events categories reported during post-op follow up 6 weeks
Arm/Group | ISB Only Adverse Events | ICG Adverse Events
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/180
Other Adverse Events (participants affected / at risk) | 5/20 | 29/180
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ISB Only Adverse Events (N=20) | ICG Adverse Events (N=180)
Reproductive system complications (Reproductive system and breast disorders) | 2 | 7 — The following were effected: Vaginal discharge Vasomotor symptoms Vaginal spotting Uterovaginal fistula Vaginal bleeding Pelvic abscess Vaginal leakage
Renal and urinary complications (Renal and urinary disorders) | 0 | 4 — The following were effected: Acute renal insufficiency Polyuria Transient right hydronephrosis Urinary retention
Wound complications (Surgical and medical procedures) | 2 | 1 — The following were effected: Wound dehiscence Wound seroma Left incisional drainage
Cellulitis (Skin and subcutaneous tissue disorders) | 1 | 5 — The following were effected: Cellulitis
Respiratory, thoracic, and pulmonary complications (Respiratory, thoracic and mediastinal disorders) | 0 | 3 — The following were effected: Pulmonary embolism Pleural effusions Pneumothorax
Cardiac complications (Cardiac disorders) | 1 | 3 — The following were effected: Cardiac complications Tachycardia Atrial fibrillation
Vascular complications (Vascular disorders) | 1 | 0 — The following were effected: Deep Vein Thrombosis
Gastrointestinal complications (Gastrointestinal disorders) | 0 | 3 — The following were effected: Small bowel obstruction
General disorders and administration site conditions (General disorders) | 1 | 4 — The following were effected: Hypotension Hypertension Lymphedema Fever
Blood and lymphatic system complications (Blood and lymphatic system disorders) | 2 | 8 — The following were effected: Leukocytosis Anemia Thrombocytopenia Neutropenia Lymphatic ascites

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes